CLINICAL TRIAL: NCT00048438
Title: Safety and Efficacy of Zemplar Capsule in Reducing Serum IPTH Levels in Chronic Kidney Disease Subjects (Three Times Weekly)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001-019
Record Dates: First submitted 2002-10-31; First posted 2002-11-04 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — paricalcitol

INTERVENTIONS:
Drug: paricalcitol

SUMMARY:
The objective of this study is to determine whether paricalcitol is safe and effective compared to placebo in reducing elevated serum PTH levels in patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Under care of physician at least 2 months (for CKD)
* Not on active Vitamin D therapy for at least 4 weeks prior
* If female:

  * Not of childbearing potential, OR
  * Practicing birth control
  * Not breastfeeding
* If taking phosphate binders, on a stable regimen at least 4 weeks prior
* For entry into Pretreatment Phase:

  * iPTH at least 120 pg/mL
  * GFR of 15-60 mL/min and no dialysis expected for at least 6 months
* For entry into Treatment Phase:

  * Average of 2 consecutive iPTH values of at least 150 pg/mL, taken at least 1 day apart (all values not less than 120 pg/mL
  * 2 consecutive corrected serum calcium levels between 8.0-10.0 mg/dL
  * 2 consecutive serum phosphorus levels of not more than 5.2 mg/mL

Exclusion Criteria:

* History of allergic reaction or sensitivity to similar drugs
* Acute Renal Failure within 12 weeks of study
* Chronic gastrointestinal disease
* Spot urine result demonstrating a urine-calcium-to-urine creatinine ratio of greater than 0.2, or a history of renal stones
* Taken aluminum-containing phosphate binders within last 12 weeks, or requires such medication for more than 3 weeks during study
* Current malignancy, or clinically significant liver disease
* Active granulomatous disease (TB, sarcoidosis, etc.)
* History of drug or alcohol abuse within 6 mos. prior
* Evidence of poor compliance with diet or medication
* Received any investigational drug or participated in any device trial within 30 days prior
* Taking maintenance calcitonin, bisphosphonates, or drugs that may affect calcium or bone metabolism (other than females on stable estrogen and/or progestin therapy)
* On glucocorticoids for a period of more than 14 days within the last 6 months
* HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68
Dates: Start 2002-02

PRIMARY OUTCOMES:
The efficacy endpoint is achievement of two consecutive > or = 30% decreases from baseline iPTH levels.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Williams, M.D., Study Director — Abbott
Locations (18):
- United States (17):
  - UCI Medical Center, Orange, California
  - Western Nephrology, Thornton, Colorado
  - Outcomes Research International, Inc., Hudson, Florida
  - Nephrology Association of South Miami, Miami, Florida
  - Tampa Bay Nephrology Associates, Tampa, Florida
  - Northwestern University Medical School, Chicago, Illinois
  - University of Missouri Health Sciences Center, Columbia, Missouri
  - Arms, Dodge, Robinson, Wilber and Crouch, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - NEA Research, Las Vegas, Nevada
  - North Shore University Hospital, Great Neck, New York
  - Mount Sinai School of Medicine, New York, New York
  - Wake Nephrology Associates, PA, Raleigh, North Carolina
  - Kidney and Hypertension Center, Cincinnati, Ohio
  - Dorn VA Hospital, Columbia, South Carolina
  - Dallas Nephrology Associates, Dallas, Texas
  - The Vancouver Clinic, Inc., P.S., Vancouver, Washington
- Jagiellonian University, Krakow, Poland